CLINICAL TRIAL: NCT02257190
Title: The Features Behind the Beneficial Effects of Interval-walking
Acronym: aIWS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2014-060
Record Dates: First submitted 2014-10-01; First posted 2014-10-06 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glycemic control; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Con) (Experimental): No exercise intervention.
  Interventions: Behavioral: Control
- Interval Walking - 3 min intervals (IW3) (Experimental): One hour of classical interval walking exercise (repeated cycles of 3 min of fast and 3 min of slow walking.
  Interventions: Behavioral: IW3
- Interval Walking - 1 min intervals (IW1) (Experimental): One hour of fast alternating interval walking exercise (repeated cycles of 3 min of fast and 3 min of slow walking
  Interventions: Behavioral: IW1

INTERVENTIONS:
Behavioral: Control — One hour of rest.
  Other Names: No exercise
  Arms: Control (Con)
Behavioral: IW3 — A one hour exercise bout with repeated cycles of 3 min of fast and 3 min of slow walking
  Other Names: 'Classical' interval walking; Interval walking - 3 min intervals
  Arms: Interval Walking - 3 min intervals (IW3)
Behavioral: IW1 — A one hour exercise bout with repeated cycles of 1 min of fast and 1 min of slow walking
  Other Names: 'Fast alternating' interval walking; Interval walking - 1 min intervals
  Arms: Interval Walking - 1 min intervals (IW1)

SUMMARY:
A single bout of Interval-Walking (IW) exercise is superior to energy-expenditure and time-duration matched Continuous Walking (CW) exercise upon improving glycemic control. The reason IW is superior is unknown.

This study will look into whether it is the larger peak intensity during IW or if it is the alternating exercise pattern that is responsible for the larger improvements seen.

Subjects with type 2 diabetes will be included in a crossover, counter-balanced, controlled study, where each subject will undergo three trials. Trials will be identical except the following interventions:

1. One hour of rest (Con)
2. One hour of classical interval walking (repeated cycles of 3 min of fast and 3 min of slow walking; IW3)
3. One hour of fast alternating interval walking (repeated cycles of 1 min of fast and 1 min of slow walking; IW1).

After the interventions subjects will undergo a standardized mixed meal tolerance test, with consecutive measurements of blood glucose, insulin and c-peptide.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Body mass index > 18 but < 40 m2/kg
* Agreement to pause antidiabetic medication from 2 days before to after each trial

Exclusion Criteria:

* Pregnancy
* Smoking
* Use of exogenous insulin
* Contraindication to increased levels of physical activity
* Evidence of thyroid, liver, lung, heart or kidney disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Within the first 4 hours after the interventions
  Glycemic control will be measured after each intervention. Subjects will receive a standardized mixed meal tolerance test (MMTT), and blood glucose values will be obtained during the test.

SECONDARY OUTCOMES:
Insulin secretion | Within the first 4 hours after the interventions
  Insulin and C-peptide will be measured during the MMTT
Insulin sensitivity | Within the first 4 hours after the interventions
  From the measurements og glucose and insulin during the MMTT, various indices of insulin sensitivity will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Karstoft, MD, PhD, Principal Investigator — Centre for Physical Activity Research, Rigshospitalet, Denmark
Locations (1):
- Center for Physical Activity Research (CFAS), Copenhagen, Denmark

REFERENCES:
- [Derived] Jakobsen I, Solomon TP, Karstoft K. The Acute Effects of Interval-Type Exercise on Glycemic Control in Type 2 Diabetes Subjects: Importance of Interval Length. A Controlled, Counterbalanced, Crossover Study. PLoS One. 2016 Oct 3;11(10):e0163562. doi: 10.1371/journal.pone.0163562. eCollection 2016. PMID 27695119